CLINICAL TRIAL: NCT05516914
Title: A Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LBL-007 in Combination With Tislelizumab in the Treatment of Malignancies
Brief Title: A Phase Ib/II Clinical Trial of LBL-007 Combined With Tislelizumab in the Treatment of Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-007-CN-004
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-03

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms | interventions — tislelizumab; Cisplatin; Gemcitabine; Injections; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-007 & Tislelizumab (Experimental): LBL-007 Injection; dose A or dose B; Q3W
  Interventions: Drug: LBL-007 Injection; Drug: Tislelizumab Injection; Drug: Cisplatin Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Docetaxel injection

INTERVENTIONS:
Drug: LBL-007 Injection — Initial dose - MTD; Q3W; intravenous infusion
  Other Names: LBL-007
Drug: Tislelizumab Injection — Initial dose; Q3W; intravenous infusion
  Other Names: Tislelizumab
Drug: Cisplatin Injection — Initial dose；Q3W; intravenous infusion
  Other Names: Cisplatin
Drug: Gemcitabine Hydrochloride for Injection — Initial dose；Q3W; intravenous infusion
  Other Names: Gemcitabine Hydrochloride
Drug: Docetaxel injection — Initial dose；Q3W; intravenous infusion
  Other Names: Docetaxel

SUMMARY:
This trial is an open and multicenter phase Ib/II clinical study, which aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, and effectiveness.

DETAILED DESCRIPTION:
This is an open, multicenter Phase Ib/II clinical trial of LBL-007 combined with Tislelizumab in the treatment of malignant tumors，which aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, and effectiveness.

The study was divided into two phases: Phase Ib (Part A): Dose escalation and PK expansion; Phase II includes: Part B, Part C, Part D, Part E, Part F, Part G, Part H. Part B ~ Part H will be designed and conducted based on the safety , tolerability and PK analysis of the Part A Study Part, after RP2D is determined, will be used for Part B ~ Part H cohort. Approximately 250-490 subjects will be enrolled (Specific sample size shall be subject to actual occurrence)

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the experimental treatment plan and visit plan, join the group voluntarily, and sign a written informed consent form;
2. Age ≥ 18 and ≤ 75 years old when signing the informed consent form, regardless of gender;
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) PS is 0~1;
4. The expected survival time is at least 12 weeks;
5. According to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1), the subjects enrolled have at least one measurable tumor lesion;
6. Subject has adequate organ and bone marrow function
7. Males with fertility and females of childbearing age are willing to take effective contraceptive measures (including abstinence, intrauterine device, various hormonal contraception, correct use of contraception from the signing of the informed consent form to 6 months after the last administration of the trial drug Sets, etc.); women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. Have received other unmarketed clinical research drugs or treatments within 4 weeks before using the research drug for the first time;
2. Those who have clinically uncontrollable pleural effusion, pericardial effusion or ascites, requiring repeated drainage or medical intervention;
3. Women during pregnancy or lactation;
4. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.
5. Patients with history of severe cardiovascular and cerebrovascular diseases.
6. Patients with active infection and currently requiring intravenous anti-infective treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy
  ORR (complete response (CR) + partial response (PR)), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST), refers to the percentage of study subjects who achieve a complete response or partial response
Dose-limiting toxicities（DLT） | DLT is defined as toxicity during the DLT observation period. The duration of DLT observation period is from the first dose to 3 weeks after the first dose
  DLT is defined as toxicity during the DLT observation period (3 weeks after the first dose).
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21days)
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles

SECONDARY OUTCOMES:
Cmax | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum serum concentration
immunogenicity | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects
Disease Control Rate(DCR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  DCR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD).
Duration of Response(DOR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  To measure duration of response
Tmax | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  After taking a single dose, Time to reach maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, Principal Investigator — Sun Yat-sen University
Locations (19):
- China (19):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital，Sun Yat-Sen University, Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The Jiangmen Central Hospital, Jiangmen, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Central People's Hospital of Zhanjinag, Zhanjiang, Guangdong
  - Guangxi Tumour Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First People's Hospital of Yu Lin, Yulin, Guangxi
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Zhejiang Cancer Hospital, Hangzhou, Hangzhou
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science And Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No